CLINICAL TRIAL: NCT04410107
Title: Short and Long Term Assessment of Lung Function, Exercise Capacity and Health-Related Quality of Life in Survivors of Severe COVID-19
Brief Title: Lung Function, Exercise Capacity and Health-Related Quality of Life After Severe COVID-19
Status: Completed | Type: Observational
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital de Clinicas de Porto Alegre (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Hospital Moinhos de Vento (Other); Federal University of Health Science of Porto Alegre (Other); Universidade de Passo Fundo (Other); Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Danilo C Berton, MD, Dr, Federal University of Rio Grande do Sul
Other Study IDs: 2020-0169
Record Dates: First submitted 2020-05-25; First posted 2020-06-01 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: Severe Acute Respiratory Syndrome Coronavirus 2; Pneumonia; Respiratory Distress Syndrome, Adult; Respiratory Function Tests; Exercise; Quality of Life
MeSH Terms: conditions — COVID-19; Pneumonia; Respiratory Distress Syndrome; Motor Activity | interventions — Respiratory Function Tests; Sports Nutritional Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe Pneumonia: Presence of fever or suspected lower respiratory infection, plus one of the following criteria:
  1) respiratory rate> 30 movements / min; 2) severe respiratory distress 3) Pulse oximetry (SpO2) ≤93% in room air; and/or 3) Pulmonary infiltrates> 50% on chest imaging within 24-48hrs of symptom onset.
  Interventions: Diagnostic Test: Lung Function tests; Diagnostic Test: Exercise capacity; Diagnostic Test: Exercise physiology; Diagnostic Test: Health-related quality of life; Diagnostic Test: Respiratory symptoms, symptoms of anxiety and depression, and post-traumatic stress screening
- Acute respiratory distress syndrome (ARDS): * Onset: acute, i.e. within 1 week of known clinical insult or new or worsening respiratory symptoms; and
  * Chest imaging (e.g. X-ray or CT scan): bilateral opacities, not fully explained by effusions, lobar/lung collapse or nodules; and
  * Origin of pulmonary edema: respiratory failure not fully explained by cardiac failure or fluid overload; and
  * Degree of hypoxemia: arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) ≤ 300 mm Hg with positive end-expiratory pressure ≥ 5 cm H2O.
  Interventions: Diagnostic Test: Lung Function tests; Diagnostic Test: Exercise capacity; Diagnostic Test: Exercise physiology; Diagnostic Test: Health-related quality of life; Diagnostic Test: Respiratory symptoms, symptoms of anxiety and depression, and post-traumatic stress screening

INTERVENTIONS:
Diagnostic Test: Lung Function tests — Spirometry before and after bronchodilator, lung volumes by body plethysmography, lung diffusion capacity of carbon monoxide (DLCO), respiratory system resistance by impulse oscillometry (IOS)
Diagnostic Test: Exercise capacity — 6-minute walk test (6MWT distance)
Diagnostic Test: Exercise physiology — Cardiopulmonary exercise test (CPET)
Diagnostic Test: Health-related quality of life — Short-Form Health Survey Questionnaire (SF-36)
Diagnostic Test: Respiratory symptoms, symptoms of anxiety and depression, and post-traumatic stress screening — 1. Adapted translation American Thoracic Society respiratory symptoms questionnaire;
  2. Beck Anxiety Inventory (BAI) and Beck's depression Inventory (BDI);
  3. Questionnaire for screening for post-traumatic stress symptoms (PTSD).

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a respiratory tract infection caused by a newly emergent coronavirus (SARS-CoV-2) that can progress to severe disease requiring hospitalization and oxygen support in around14% of the cases and 5% require admission in intensive care unit. The medium and long-term impact in survivors of severe COVID-19 on lung function, exercise capacity and health-related quality of life remains to be determined.

DETAILED DESCRIPTION:
Background: Coronavirus disease 2019 (COVID-19) is a respiratory tract infection caused by a newly emergent coronavirus (severe acute respiratory syndrome coronavirus 2; SARS-CoV-2) that was first recognized in Wuhan, China, in December 2019. Currently, this infection reached pandemic levels causing serious diseases in 14% of cases and the potential to progress to acute respiratory distress syndrome (ARDS) with the need for invasive ventilatory support and prolonged hospitalization in intensive care units (ICU). The overall lethality is 2% and the lethality of cases admitted to the ICU varies from 26 to 50%. The medium and long-term impact in survivors of severe COVID-19 on lung function, exercise capacity and health related quality of life (HRQoL) remains to be determined.

Aims: To evaluate the early (Visit1: 2-6 months after acute disease) and late (Visit 2: 9-15 months and Visit 3: 18-24 months) effects of severe acute respiratory syndrome on lung function, exercise capacity, respiratory symptoms and HRQoL in patients with confirmed diagnosis of SARS-CoV-2 infection.

Material and methods: Prospective cohort of subjects with laboratory confirmed severe COVID-19 (respiratory rate> 30 breaths/ min; severe respiratory distress; oxyhemoglobin saturation in room air ≤93% or pulmonary involvement> 50% in chest images). Participants will perform spirometry before and after bronchodilator, lung volumes by body plethysmography, lung diffusion capacity of carbon monoxide, respiratory system resistance by impulse oscillometry and 6-minute walk test (6MWT) after 2-6 months (Visit 1) , 9-15 months (Visit 2), and 18-24 months (Visit 3) of severe COVID-19. When abnormalities in these pulmonary function tests and/or 6MWT were detected, a cardiopulmonary exercise test will be performed. Clinical, laboratory and chest image data during the severe COVID-19 hospitalization will be obtained from medical records.

The minimum sample size was estimated as 134 participants to assess at least 5 independent factors to predict lung function, HRQoL and exercise capacity at the early assessment. Notwithstanding, the investigators plan to invite to participate all survivors of severe COVID-19 admitted in hospitals of the state of Rio Grande do Sul (Brazil).

ELIGIBILITY:
Inclusion Criteria:

* Previous laboratory confirmation of SARS-Cov-2 infection defined as a positive result of reverse polymerase-transcriptase chain reaction test in real-time of a sample taken by nasal and/or pharyngeal swab; and
* Severe pneumonia defined by the presence of fever or suspected lower respiratory infection, plus one of the following criteria: respiratory rate> 30 movements/min; severe respiratory distress; SpO2≤93% in room air; or pulmonary infiltrates>50% on chest imaging within 24-48hrs of acute symptoms onset; and/or
* Acute respiratory distress syndrome (ARDS) defined according to COVID-19 operational management guide of World Health Organization and classified as mild (200 mmHg <PaO2 / FiO2 ≤ 300 mmHg), moderate (100 mmHg <PaO2 / FiO2 ≤ 200 mmHg) or severe (PaO2 / FiO2 ≤ 100 mmHg). When the PaO2 is not available, SpO2 / FiO2 ≤ 315 suggests ARDS.

Exclusion Criteria:

* Lack of clinical stability for 2 months before inclusion (including those who remain hospitalized);
* Active respiratory tract infection (of any cause); or
* Any clinical condition that prevents the performance of the study procedures.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects that survived severe COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2020-05-15 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in the first second/forced vital capacity | 6 months
  ratio obtained from measured values during spirometry
Total lung capacity | 6 months
  obtained from plethysmography (% of predicted)
Lung diffusion capacity for carbon monoxide | 6 months
  obtained from single-breathe maneuver (% of predicted)
6-minute walk test distance | 6 months
  distance walked during the test (m)
Short-form 36 questionnaire (SF-36) | 6 months
  scores range between 0 and 100 with higher scores indicating a better HRQoL

SECONDARY OUTCOMES:
Forced expiratory volume in the first second/forced vital capacity | 12 and 24 months
  ratio obtained from measured values during spirometry
Forced vital capacity | 6, 12 and 24 months
  % of predicted
Residual volume/total lung capacity | 6, 12 and 24 months
  ratio obtained from measured values during plethysmography
Inspiratory capacity/total lung capacity | 6, 12 and 24 months
  ratio obtained from measured values during plethysmography
Airway resistance (Raw) | 6, 12 and 24 months
  obtained from body plethysmography
Lung diffusion capacity for carbon monoxide | 12 and 24 months
  obtained from single-breathe maneuver (% of predicted)
Resistance at 20Hz and 5Hz (R5-R20) | 6, 12 and 24 months
  obtained from Impulse oscillometry
Reactance at 5Hz (X5) | 6, 12 and 24 months
  obtained from Impulse oscillometry
Resonant frequency (Fres) | 6, 12 and 24 months
  obtained from Impulse oscillometry
Reactance area (AХ) | 6, 12 and 24 months
  obtained from Impulse oscillometry
6-minute walk test distance | 12 and 24 months
  distance walked during the test (m)
Pulse oximetry (SpO2) at rest | 6, 12 and 24 months
  before 6-minute walk test
Pulse oximetry (SpO2) during exercise | 6, 12 and 24 months
  at the end of 6-minute walk test
Respiratory symptoms adapted from American Thoracic Society Questionnaire | 6, 12 and 24 months
  descriptive/qualitative questionnaire
Short-form 36 questionnaire (SF-36) | 12 and 24 months
  scores range between 0 and 100 with higher scores indicating a better HRQoL
Oxygen uptake at peak exercise | 6, 12 and 24 months
  from incremental Cardiopulmonary exercise test (% of predicted)
Minute-ventilation/carbon dioxide output during exercise | 6, 12 and 24 months
  from incremental Cardiopulmonary exercise test (L/L)
Dyspnea during exercise | 6, 12 and 24 months
  from incremental Cardiopulmonary exercise test (measured with 10-point categorical Borg scale)
Inspiratory capacity during exercise | 6, 12 and 24 months
  from incremental Cardiopulmonary exercise test (L and % of predicted)
Beck Anxiety Inventory (BAI) | 6, 12 and 24 months
  total score ranges from 0 to 63; higher score indicating higher anxiety
Beck Depression Inventory (BDI) | 6, 12 and 24 months
  total scores ranges from 0 to 63; higher score is worse
Post-traumatic stress symptoms questionnaire | 6, 12 and 24 months
  17-item, 5 likert-scale each item; higher score indicating more symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Danilo C Berton, Dr, Principal Investigator — Universidade Federal do Rio Grande do Sul/Hospital de Clínicas de Porto Alegre
Locations (5):
- Brazil (5):
  - Universidade de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre/Universidade Federal do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Univesidade de Ciências da Saúde de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceição, Porto Alegre, Rio Grande do Sul

REFERENCES:
- [Derived] Benedetto IG, Silva RMCD, Hetzel GM, Viana GDS, Guimaraes AR, Folador L, Brentano VB, Garcia TS, Ribeiro SP, Dalcin PTR, Gazzana MB, Berton DC. Impact of impaired pulmonary function on clinical outcomes in survivors of severe COVID-19 without pre-existing respiratory disease. J Bras Pneumol. 2023 May 26;49(3):e20220452. doi: 10.36416/1806-3756/e20220452. eCollection 2023. PMID 37255163